CLINICAL TRIAL: NCT02101034
Title: Phase I/II Trial of the Addition of PD 0332991 to Cetuximab in Patients With Incurable SCCHN
Brief Title: PD 0332991 and Cetuximab in Patients With Incurable SCCHN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201404139
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Results first posted 2021-06-11 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase I: Dose Level 1 (Experimental): PD 0332991 will be administered on Days 1 through 21 of each 28 day cycle.
  Cetuximab will be administered intravenously on a weekly schedule. The first dose will be 400 mg/m2. The remaining weekly dose will be 250 mg/m2. Participants will continue to receive weekly cetuximab at 250 mg/m2 for the duration of their participation on study.
  Interventions: Biological: Cetuximab; Drug: PD 0332991
- Phase I: Dose Level 2 (Experimental): PD 0332991 will be administered on Days 1 through 21 of each 28 day cycle.
  Cetuximab will be administered intravenously on a weekly schedule. The first dose will be 400 mg/m2. The remaining weekly dose will be 250 mg/m2. Participants will continue to receive weekly cetuximab at 250 mg/m2 for the duration of their participation on study.
  Interventions: Biological: Cetuximab; Drug: PD 0332991
- Phase II Arm 1: Platin-Resistant HPV-Unrelated SCCHN (Experimental): PD 0332991 will be administered on Days 1 through 21 of each 28 day cycle.
  Cetuximab will be administered intravenously on a weekly schedule. The first dose will be 400 mg/m2. The remaining weekly dose will be 250 mg/m2. Participants will continue to receive weekly cetuximab at 250 mg/m2 for the duration of their participation on study.
  Interventions: Biological: Cetuximab; Drug: PD 0332991
- Phase II Arm 2: Cetuximab-Resistant HPV-Unrelated SCCHN (Experimental): PD 0332991 will be administered on Days 1 through 21 of each 28 day cycle.
  Cetuximab will be administered intravenously on a weekly schedule. The first dose will be 400 mg/m2. The remaining weekly dose will be 250 mg/m2. Participants will continue to receive weekly cetuximab at 250 mg/m2 for the duration of their participation on study.
  Interventions: Biological: Cetuximab; Drug: PD 0332991
- Phase II Arm 3: (Experimental): PD 0332991 will be administered on Days 1 through 21 of each 28 day cycle.
  Cetuximab will be administered intravenously on a weekly schedule. The first dose will be 400 mg/m2. The remaining weekly dose will be 250 mg/m2. Participants will continue to receive weekly cetuximab at 250 mg/m2 for the duration of their participation on study.
  Interventions: Biological: Cetuximab; Drug: PD 0332991

INTERVENTIONS:
Biological: Cetuximab
  Other Names: Erbitux®
Drug: PD 0332991
  Other Names: palbociclib

SUMMARY:
The purpose of this Phase I/II study is to define the maximum tolerated dose of PD 0332991 given with cetuximab and evaluated the side effects of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of squamous cell carcinoma of the head and neck.
* Disease must be considered incurable. Incurable is defined as metastatic disease or a local or regional recurrence in a previously irradiated site that is unresectable (or patient declines resection).
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥10 mm with CT scan, as ≥20 mm by chest x-ray, or ≥10 mm with calipers by clinical exam. (Phase I only: patients without measurable disease by RECIST 1.1 criteria but with evaluable disease by imaging or physical exam will be eligible as well.)
* Phase I only: any (or no) prior therapy for metastatic disease is allowed, including cetuximab. If a patient has not received prior standard therapy, s/he must have been offered and refused prior standard therapy.
* Phase II only:

  * Arm 1: disease progression after at least one cycle of prior treatment with cisplatin or carboplatin for incurable disease. Prior treatment with cetuximab for incurable disease is not permitted.
  * Arms 2 and 3: disease progression after at least one cycle of treatment with cetuximab for incurable disease.
* Phase II only: at least one line of prior therapy for incurable disease.
* Phase II only:

  * Arms1 and 2: disease must be determined to be HPV-unrelated. HPV-unrelated SCCHN is defined as either p16-negative OPSCC or non-OPSCC (larynx, hypopharynx, oral cavity) or p16-negative unknown primary SCC presenting with a level 2 or 3 neck node. p16 will be assessed by IHC; a specimen showing any staining will be considered p16-positive.
  * Arm 3: disease must be HPV-related SCCHN (defined as OPSCC or unknown primary presenting with a neck mass that is either p16 positive or HPV ISH or PCR positive).
* Minimum of 14 days elapsed since the end of any prior therapy.
* At least 18 years of age.
* Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCI CTCAE version 4.0 Grade ≤ 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion)
* ECOG performance status ≤ 2
* Adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500 mm3
  * Platelets ≥ 100,000 mm3
  * Hemoglobin > 9 g/dL
  * Total bilirubin ≤ 1.5 x IULN except in the case of patients with Gilbert's disease
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 x IULN for patients without liver metastases and ≤ 5.0 x IULN for patients with liver metastases
  * Alkaline phosphatase ≤ 2.5 x IULN for patients without bone metastases and ≤ 5.0 x IULN for patients with bone metastases
  * Serum creatinine ≤ 1.5 x IULN OR calculated creatinine clearance ≥ 50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Baseline corrected QT interval (QTc) < 480 ms.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Available archival tumor tissue for the proposed correlative studies.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Phase II, Arm 1 only: prior treatment with cetuximab.
* Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCI CTCAE version 4.0 Grade ≤ 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator´s discretion)
* A history of other malignancy ≤ 1 year previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only, carcinoma in situ of the cervix, or synchronous H&N primaries.
* Currently receiving any other investigational agents.
* Patient must not have a history of or clinical evidence of central nervous system metastases or leptomeningeal carcinomatosis, except for individuals who have had previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medications (with the exception of Keppra) for 1 month prior to first dose of PD 0332991.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to PD 0332991, cetuximab, or other agents used in the study.
* Treated within the last 7 days prior to Day 1 of protocol therapy with:

  * Food or drugs that are known to be CYP3A4 inhibitors (e.g. grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, clarithromycin, telithromycin, indinavir, ritonavir, nelfinavir, atazanavir, amprenavir, nefazodone, diltiazem, and delavirdine) or inducers (i.e. dexamethasone, glucocorticoids, progesterone, rifampin, phenobarbital, St. John's wort).
  * Drugs that are known to prolong the QT interval.
  * Drugs that are proton pump inhibitors.
* Uncontrolled electrolyte disorders that can compound the effects of a QTc-prolonging drug (e.g., hypocalcemia, hypokalemia, hypomagnesemia)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 28 days of study entry. Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraceptive during the period of the trial and for at least 90 days after completion of treatment. The decision of effective contraception will be based on the judgment of the principal investigator or a designated associate.
* Phase I and Arm 1 of Phase II: Known HIV-positivity and on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with PD 0332991. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Arms 2 and 3 of Phase II: patients with HIV infection and antiretroviral therapy are not excluded, as there are no pharmacokinetic tests being performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-06-17 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2023-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (5):
- United States (5):
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Kansas, Westwood, Kansas
  - University of Michigan Health System, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adkins D, Ley J, Neupane P, Worden F, Sacco AG, Palka K, Grilley-Olson JE, Maggiore R, Salama NN, Trinkaus K, Van Tine BA, Steuer CE, Saba NF, Oppelt P. Palbociclib and cetuximab in platinum-resistant and in cetuximab-resistant human papillomavirus-unrelated head and neck cancer: a multicentre, multigroup, phase 2 trial. Lancet Oncol. 2019 Sep;20(9):1295-1305. doi: 10.1016/S1470-2045(19)30405-X. Epub 2019 Jul 24. PMID 31351869
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Dose Level 1: PD 0332991 100 mg per day will be administered on Days 1 through 21 of each 28 day cycle.
  Cetuximab will be administered intravenously on a weekly schedule. The first dose will be 400 mg/m2. The remaining weekly dose will be 250 mg/m2. Participants will continue to receive weekly cetuximab at 250 mg/m2 for the duration of their participation on study.
- Phase I: Dose Level 2; Phase II Arm 1: Platin-Resistant HPV-Unrelated SCCHN; Phase II Arm 2: Cetuximab-Resistant HPV-Unrelated SCCHN; Phase II Arm 3:: PD 0332991 125 mg per day will be administered on Days 1 through 21 of each 28 day cycle.
  Cetuximab will be administered intravenously on a weekly schedule. The first dose will be 400 mg/m2. The remaining weekly dose will be 250 mg/m2. Participants will continue to receive weekly cetuximab at 250 mg/m2 for the duration of their participation on study.
Period: Overall Study
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II Arm 1: Platin-Resistant HPV-Unrelated SCCHN | Phase II Arm 2: Cetuximab-Resistant HPV-Unrelated SCCHN | Phase II Arm 3:
Started | 3 | 6 | 31 | 32 | 24
Completed | 3 | 6 | 30 | 32 | 24
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Enrolled but did not start treatment | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II Arm 1: Platin-Resistant HPV-Unrelated SCCHN | Phase II Arm 2: Cetuximab-Resistant HPV-Unrelated SCCHN | Phase II Arm 3: | Total
Number analyzed (Participants) | 3 | 6 | 31 | 32 | 24 | 96
Age, Continuous [Median (Full Range); unit: years] | 62 [57 to 78] | 61 [37 to 64] | 64 [26 to 84] | 64 [49 to 77] | 66 [45 to 71] | 63 [26 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 7 | 11 | 2 | 22
  Male | 3 | 4 | 24 | 21 | 22 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 3 | 6 | 30 | 30 | 23 | 92
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 7 | 7 | 0 | 16
  White | 3 | 3 | 23 | 24 | 24 | 77
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 31 | 32 | 24 | 96

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Maximum Tolerated Dose (MTD)
Description: MTD is the dose level (DL) immediately below the DL at which 2 patients of a cohort experience dose limiting toxicity (DLT) in the 1st cycle (DLTs) Hematologic DLT is any of the below that occur during the 1st cycle that are possibly, probably, or definitely related to the treatment grade 4 neutropenia ≥7 days grade 4 infection with grade 3/4 neutropenia grade 4 thrombocytopenia with life-threatening bleeding treatment held for >14 days due to hematologic toxicity febrile neutropenia with temperature >=38.5°C
  Non-hematologic DLT is any possibly, probably, or definitely related grade 3 or 4 non-hematologic toxicity that occurs during the 1st except for suboptimally treated grade 3 or 4 nausea, vomiting, diarrhea, anorexia, or lymphopenia grade 3 metabolic abnormalities (limited to potassium, magnesium, and calcium) any hypersensitivity/infusion reaction or acneiform rash due to cetuximab treatment held for >14 days due to non-hematologic toxicity
Time Frame: 6 months (estimated completion of Phase I)
Population: Only Phase I participants were evaluable for this outcome measure.
Measure: Number; unit: mg
Groups:
- Phase I: Dose Level 1 and Dose Level 2: * PD 0332991 will be administered on Days 1 through 21 of each 28 day cycle.
  * Dose Level 1 PD 0332991 100 mg per day
  * Dose Level 2 PD 0332991 125 mg per day
  Cetuximab will be administered intravenously on a weekly schedule. The first dose will be 400 mg/m2. The remaining weekly dose will be 250 mg/m2. Participants will continue to receive weekly cetuximab at 250 mg/m2 for the duration of their participation on study.
Arm/Group | Phase I: Dose Level 1 and Dose Level 2 | Phase II Arm 1: Platin-Resistant HPV-Unrelated SCCHN | Phase II Arm 2: Cetuximab-Resistant HPV-Unrelated SCCHN | Phase II Arm 3:
Number analyzed (Participants) | 9 | 0 | 0 | 0
mg | NA — None of the nine participants enrolled in the Phase I portion of the study experienced a dose-limiting toxicity. A MTD of palbociclib was not reached. |  |  |

2. Primary Outcome: Phase II: Efficacy as Measured by Overall Response Rate
Description: Tumor measurements will be collected at baseline, end of every even numbered cycles, and end of treatment.
  Measured by overall response rate (ORR=CR+PR) defined by RECIST criteria
  Best overall response is the best response recorded from the start of treatment until disease progression/recurrence
  Complete Response (CR) is defined as disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  Partial Response (PR) is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters
Time Frame: End of treatment (estimated to be 12 months)
Population: Phase I participants were excluded from this outcome measure. 2 participants in Phase II Arm 1 were not evaluable due to early death and inability to measure the target lesion on the post-treatment non-contrast CT scan. 5 participants in Phase II Arm 2 were not evaluable due to comorbidity-related death (N=2), patient withdrawal (N=2), and non-treatment related adverse event (N=1).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II Arm 1: Platin-Resistant HPV-Unrelated SCCHN | Phase II Arm 2: Cetuximab-Resistant HPV-Unrelated SCCHN | Phase II Arm 3:
Number analyzed (Participants) | 0 | 0 | 28 | 27 | 24
Participants |  |  | 11 | 5 | 1

3. Secondary Outcome: Phase I: Most Frequent Adverse Events
Description: Assessed by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: Up to 30 days following completion of treatment (estimated to be 13 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2
Number analyzed (Participants) | 3 | 6
Participants
  Grades 1-2 Neutropenia | 1 | 2
  Grade 3 Neutropenia | 1 | 2
  Grades 1-2 Anemia | 2 | 6
  Grade 3 Anemia | 1 | 0
  Grades 1-2 Thrombocytopenia | 1 | 3
  Grade 3 Thrombocytopenia | 1 | 0
  Grades 1-2 Fatigue | 2 | 3
  Grade 3 Fatigue | 0 | 0
  Grades 1-2 Nausea | 0 | 2
  Grade 3 Nausea | 0 | 0
  Grade 1-2 Vomiting | 0 | 1
  Grade 3 Vomiting | 0 | 0
  Grade 1-2 Diarrhea | 1 | 1
  Grade 3 Diarrhea | 0 | 0
  Grade 1-2 Infusion Reaction | 0 | 1
  Grade 3 Infusion Reaction | 0 | 0
  Grade 1-2 Acneiform Rash | 2 | 5
  Grade 3 Acneiform Rash | 0 | 0
  Grade 1-2 Hypomagnesemia | 1 | 2
  Grade 3 Hypomagnesemia | 1 | 0

4. Secondary Outcome: Phase II: PD 0332991 Related Adverse Events Occurring in 10% or More of Participants and All Grade 3-5 Adverse Events
Description: Assessed by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: Up to 30 days following completion of treatment (estimated to be 13 months)
Population: All arms of the Phase II Portion of the study were combined for this outcome measure as the treatment received was the same for each arm.
Measure: Count of Participants; unit: Participants
Groups:
- Phase II Arm 1, Arm 2, and Arm 3: PD 0332991 125 mg per day will be administered on Days 1 through 21 of each 28 day cycle.
  Cetuximab will be administered intravenously on a weekly schedule. The first dose will be 400 mg/m2. The remaining weekly dose will be 250 mg/m2. Participants will continue to receive weekly cetuximab at 250 mg/m2 for the duration of their participation on study.
Arm/Group | Phase II Arm 1, Arm 2, and Arm 3
Number analyzed (Participants) | 86
Participants
  Grades 1-2 platelet count decreased | 50
  Grades 3-5 platelet count decreased | 11
  Grades 1-2 neutrophil count decreased | 28
  Grades 3-5 neutrophil count decreased | 29
  Grades 1-2 white blood cell count decreased | 43
  Grades 3-5 white blood cell count decreased | 24
  Grades 1-2 electrocardiogram QT corrected interval prolonged | 6
  Grades 3-5 electrocardiogram QT corrected interval prolonged | 1

5. Secondary Outcome: Phase II: Cetuximab Related Adverse Events Occurring in 10% or More of Participants and All Grade 3-5 Adverse Events
Description: Assessed by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: Up to 30 days following completion of treatment (estimated to be 13 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Arm 1, Arm 2, and Arm 3
Number analyzed (Participants) | 86
Participants
  Grades 1-2 acneiform rash | 60
  Grades 3-5 acneiform rash | 0
  Grades 1-2 hypomagnesemia | 23
  Grades 3-5 hypomagnesemia | 1

6. Secondary Outcome: Phase II: Adverse Events Occurring in 10% or More of Participants and All Grade 3-5 Adverse Events
Description: Assessed by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: Up to 30 days following completion of treatment (estimated to be 13 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- Phase II: Arm 1, Arm 2, and Arm 3: PD 0332991 125 mg per day will be administered on Days 1 through 21 of each 28 day cycle.
  Cetuximab will be administered intravenously on a weekly schedule. The first dose will be 400 mg/m2. The remaining weekly dose will be 250 mg/m2. Participants will continue to receive weekly cetuximab at 250 mg/m2 for the duration of their participation on study.
Arm/Group | Phase II: Arm 1, Arm 2, and Arm 3
Number analyzed (Participants) | 86
Participants
  Grades 1-2 fatigue | 48
  Grades 3-5 fatigue | 8
  Grades 1-2 hypoalbuminemia | 37
  Grades 3-5 hypoalbuminemia | 3
  Grades 1-2 anemia | 44
  Grades 3-5 anemia | 20
  Grades 1-2 hyponatremia | 30
  Grades 3-5 hyponatremia | 1
  Grades 1-2 hypertension | 24
  Grades 3-5 hypertension | 3
  Grades 1-2 nausea | 30
  Grades 3-5 nausea | 3
  Grades 1-2 dysphagia | 30
  Grades 3-5 dysphagia | 6
  Grades 1-2 dyspnea | 29
  Grades 3-5 dyspnea | 5
  Grades 1-2 hypocalcemia | 19
  Grades 3-5 hypocalcemia | 4
  Grades 1-2 lymphocyte count decreased | 19
  Grades 3-5 lymphocyte count decreased | 22
  Grades 1-2 diarrhea | 21
  Grades 3-5 diarrhea | 2
  Grades 1-2 weight loss | 24
  Grades 3-5 weight loss | 6
  Grades 1-2 AST increased | 22
  Grades 3-5 AST increased | 0
  Grades 1-2 tumor pain | 18
  Grades 3-5 tumor pain | 3
  Grades 1-2 constipation | 15
  Grades 3-5 constipation | 0
  Grades 1-2 cough | 21
  Grades 3-5 cough | 0
  Grades 1-2 anorexia | 21
  Grades 3-5 anorexia | 3
  Grades 1-2 vomiting | 17
  Grades 3-5 vomiting | 2
  Grades 1-2 dry mouth | 13
  Grades 3-5 dry mouth | 0
  Grades 1-2 sinus tachycardia | 12
  Grades 3-5 sinus tachycardia | 0
  Grades 1-2 alkaline phosphatase increased | 12
  Grades 3-5 alkaline phosphatase increased | 0
  Grades 1-2 hypokalemia | 12
  Grades 3-4 hypokalemia | 11
  Grades 1-2 hyperglycemia | 11
  Grades 3-5 hyperglycemia | 11
  Grades 1-2 hypernatremia | 16
  Grades 3-5 hypernatremia | 1
  Grades 1-2 fever | 12
  Grades 3-5 fever | 1
  Grades 1-2 dizziness | 9
  Grades 3-5 dizziness | 2
  Grades 1-2 hypercalcemia | 9
  Grades 3-5 hypercalcemia | 1
  Grades 1-2 dry skin | 18
  Grades 3-5 dry skin | 1
  Grades 1-2 dehydration | 8
  Grades 3-5 dehydration | 2
  Grades 1-2 hypotension | 8
  Grades 3-5 hypotension | 1
  Grades 1-2 creatinine increased | 12
  Grades 3-5 creatinine increased | 1
  Grades 1-2 trismus | 7
  Grades 3-5 trismus | 1
  Grades 1-2 elevated INR | 6
  Grades 3-5 elevated INR | 1
  Grades 1-2 dysarthria | 5
  Grades 3-5 dysarthria | 1
  Grades 1-2 hypophosphatemia | 3
  Grades 3-5 hypophosphatemia | 8
  Grades 1-2 lung infection | 1
  Grades 3-5 lung infection | 8
  Grades 1-2 febrile neutropenia | 0
  Grades 3-5 febrile neutropenia | 2
  Grade 1-2 abdominal pain | 0
  Grades 3-5 abdominal pain | 2
  Grades 1-2 colitis | 0
  Grades 3-5 colitis | 1
  Grades 1-2 tumor hemorrhage | 0
  Grades 3-5 tumor hemorrhage | 2
  Grades 1-2 hematuria | 0
  Grades 3-5 hematuria | 1
  Grades 1-2 duodenal ulcer | 0
  Grades 3-5 duodenal ulcer | 1
  Grades 1-2 esophageal fistula | 0
  Grades 3-5 esophageal fistula | 1
  Grades 1-2 oral cavity fistula | 0
  Grades 3-5 oral cavity fistula | 1
  Grades 1-2 sepsis | 0
  Grades 3-5 sepsis | 7
  Grades 1-2 duodenal perforation | 0
  Grades 3-5 duodenal perforation | 1
  Grades 1-2 skin infection | 0
  Grades 3-5 skin infection | 4
  Grades 1-2 tracheitis | 0
  Grades 3-5 tracheitis | 1
  Grades 1-2 aspiration | 0
  Grades 3-5 aspiration | 1
  Grades 1-2 pleural effusion | 0
  Grades 3-5 pleural effusion | 1
  Grades 1-2 pneumothorax | 0
  Grades 3-5 pneumothorax | 1
  Grades 1-2 catheter-related infection | 0
  Grades 3-5 catheter-related infection | 1
  Grades 1-2 jejunal obstruction | 0
  Grades 3-5 jejunal obstruction | 1
  Grades 1-2 mucositis oral | 4
  Grades 3-5 mucositis oral | 2
  Grades 1-2 oral hemorrhage | 0
  Grades 3-5 oral hemorrhage | 1
  Grade 5 death, not otherwise specified | 3
  Grades 1-2 infusion-related reaction | 0
  Grades 3-5 infusion-related reaction | 1
  Grades 1-2 urinary tract infection | 0
  Grades 3-5 urinary tract infection | 2
  Grades 1-2 respiratory failure | 0
  Grades 3-5 respiratory failure | 2
  Grades 1-2 hypothyroidism | 5
  Grades 3-5 hypothyroidism | 0
  Grades 1-2 edema face | 2
  Grades 3-5 edema face | 1
  Grades 1-2 non-cardiac chest pain | 2
  Grades 3-5 non-cardiac chest pain | 1
  Grades 1-2 pancreatitis | 0
  Grades 3-5 pancreatitis | 1
  Grades 1-2 encephalopathy | 0
  Grades 3-5 encephalopathy | 1
  Grades 1-2 acute kidney injury | 0
  Grades 3-5 acute kidney injury | 1
  Grades 1-2 proteinuria | 0
  Grades 3-5 proteinuria | 1
  Grades 1-2 thromboembolic event | 0
  Grades 3-5 thromboembolic event | 1

7. Secondary Outcome: Phase II: Progression Free Survival (PFS)
Description: Participants were followed every 2 months for up to 5 years or until death, whichever occurs first.
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II Arm 1: Platin-Resistant HPV-Unrelated SCCHN | Phase II Arm 2: Cetuximab-Resistant HPV-Unrelated SCCHN | Phase II Arm 3:
Number analyzed (Participants) | 30 | 32 | 24
months | 5.72 [3.97 to 7.93] | 3.75 [2.93 to 4.37] | 1.82 [1.77 to 2.10]

8. Secondary Outcome: Phase II: Overall Survival (OS)
Description: Participants were followed every 2 months for up to 5 years or until death, whichever occurs first.
  Overall survival is measured from time of diagnosis to time of death.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II Arm 1: Platin-Resistant HPV-Unrelated SCCHN | Phase II Arm 2: Cetuximab-Resistant HPV-Unrelated SCCHN | Phase II Arm 3:
Number analyzed (Participants) | 30 | 32 | 24
months | 9.75 [5.57 to 15.53] | 7.00 [4.97 to 9.37] | 9.32 [4.39 to 18.35]

9. Secondary Outcome: Phase II: Duration of Response
Description: Duration of overall response is measured from the time measurement criteria are met for CR or PR until the first date that recurrent or progressive disease is objectively documented.
Time Frame: Completion of treatment (estimated to be 12 months)
Population: Phase I participants were not evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II Arm 1: Platin-Resistant HPV-Unrelated SCCHN | Phase II Arm 2: Cetuximab-Resistant HPV-Unrelated SCCHN | Phase II Arm 3:
Number analyzed (Participants) | 0 | 0 | 11 | 5 | 1
months |  |  | 4.0 [1.8 to 5.6] | 6.0 [2.0 to 15.5] | 4.0

ADVERSE EVENTS:
Time Frame: Adverse events were followed from start of study treatment until 30 days following the last day of study treatment, up to approximately 13 months. All-Cause Morality was assessed from start of study treatment up to 5 years.
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II Arm 1: Platin-Resistant HPV-Unrelated SCCHN | Phase II Arm 2: Cetuximab-Resistant HPV-Unrelated SCCHN | Phase II Arm 3:
All-Cause Mortality (participants affected / at risk) | 3/3 | 6/6 | 26/30 | 19/32 | 15/24
Serious Adverse Events (participants affected / at risk) | 2/3 | 4/6 | 21/30 | 16/32 | 9/24
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 30/30 | 32/32 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Dose Level 1 (N=3) | Phase I: Dose Level 2 (N=6) | Phase II Arm 1: Platin-Resistant HPV-Unrelated SCCHN (N=30) | Phase II Arm 2: Cetuximab-Resistant HPV-Unrelated SCCHN (N=32) | Phase II Arm 3: (N=24)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Esophageal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Jejunal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausa (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Oral cavity fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Death NOS (General disorders) | 0 | 0 | 3 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 1 | 0 | 0
Failure to thrive (General disorders) | 0 | 0 | 1 | 0 | 0
Fall (General disorders) | 0 | 0 | 2 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0 | 0
Fever (General disorders) | 0 | 0 | 1 | 1 | 2
Infusion related reaction (General disorders) | 0 | 0 | 1 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 8 | 3 | 3
Meningitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 2 | 3 | 1
Skin infection (Infections and infestations) | 0 | 1 | 2 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Intestinal stoma leak (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Facial muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Dose Level 1 (N=3) | Phase I: Dose Level 2 (N=6) | Phase II Arm 1: Platin-Resistant HPV-Unrelated SCCHN (N=30) | Phase II Arm 2: Cetuximab-Resistant HPV-Unrelated SCCHN (N=32) | Phase II Arm 3: (N=24)
Anemia (Blood and lymphatic system disorders) | 3 | 6 | 30 | 24 | 17
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Constrictive pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 3 | 1 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 20 | 12 | 4
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 0
Hearing imparied (Ear and labyrinth disorders) | 0 | 0 | 5 | 1 | 2
Otorrhea (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 1 | 0
Hypoparathyroidism (Endocrine disorders) | 0 | 0 | 5 | 0 | 0
Hypothrydodism (Endocrine disorders) | 0 | 0 | 0 | 4 | 5
Blurred vision (Eye disorders) | 0 | 0 | 2 | 1 | 0
Conjuctivitis (Eye disorders) | 0 | 0 | 3 | 2 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye discomfort (Eye disorders) | 0 | 0 | 1 | 0 | 0
Melanocytic nevus (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 4
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 9 | 6 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 12 | 10 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 3 | 18 | 13 | 10
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 3 | 19 | 13 | 8
Esophageal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 5
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Hypersalivation (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0
Mouth sores (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 10 | 5 | 5
Nausea (Gastrointestinal disorders) | 0 | 2 | 10 | 18 | 7
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oral bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Oral cavity fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 2 | 2 | 1 | 2 | 3
Rectal bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Sore tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 5 | 10 | 3
Chills (General disorders) | 0 | 0 | 8 | 5 | 3
Edema face (General disorders) | 0 | 0 | 4 | 4 | 3
Edema limbs (General disorders) | 0 | 0 | 6 | 2 | 2
Facial pain (General disorders) | 0 | 0 | 2 | 0 | 2
Fall (General disorders) | 0 | 1 | 4 | 3 | 2
Fatigue (General disorders) | 2 | 3 | 26 | 18 | 17
Fever (General disorders) | 0 | 0 | 6 | 3 | 1
Flu like symptoms (General disorders) | 0 | 1 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 1 | 0 | 0 | 0
Infusion related reaction (General disorders) | 0 | 1 | 3 | 0 | 2
Irritability (General disorders) | 0 | 0 | 1 | 0 | 0
Localized edema (General disorders) | 0 | 0 | 2 | 1 | 0
Localized edema (General disorders) | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 6 | 3 | 1
Neck edema (General disorders) | 0 | 0 | 2 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 5 | 0 | 3
Pain (General disorders) | 0 | 0 | 2 | 1 | 1
Pain in extremity (General disorders) | 0 | 0 | 2 | 0 | 1
Restless leg (General disorders) | 0 | 0 | 0 | 0 | 1
Upper back edema (General disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Bone infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bronchial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpertic blepharitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Nail infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 1 | 12 | 5 | 5
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 6 | 3 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0 | 2 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Hand wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Intestinal stoma leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skin ulceration (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 0 | 1
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1 | 5 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 7 | 1 | 2
Alkaline phosphatase increased (Investigations) | 0 | 1 | 7 | 6 | 7
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 10 | 6 | 6
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0
CPK increased (Investigations) | 0 | 0 | 1 | 0 | 0
Cardiac troponin I increased (Investigations) | 0 | 0 | 3 | 0 | 0
Cholesterol high (Investigations) | 0 | 0 | 1 | 1 | 1
Creatinine increased (Investigations) | 1 | 2 | 8 | 2 | 5
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 10 | 2 | 1
GGT increased (Investigations) | 0 | 0 | 1 | 0 | 0
INR increased (Investigations) | 1 | 2 | 15 | 7 | 4
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 3 | 6 | 28 | 14 | 19
Neutrophil count decreased (Investigations) | 2 | 4 | 26 | 18 | 14
Platelet count decreased (Investigations) | 2 | 3 | 23 | 23 | 16
Weight loss (Investigations) | 0 | 0 | 15 | 9 | 8
White blood cell decreased (Investigations) | 2 | 6 | 26 | 23 | 19
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 4 | 3 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 17 | 6 | 7
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 5 | 5 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 8 | 4 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 10 | 11 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 3 | 1
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 6 | 5 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 3 | 20 | 15 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 4 | 17 | 7 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 5 | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 13 | 9 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 2 | 13 | 10 | 5
Hyponatremia (Metabolism and nutrition disorders) | 1 | 4 | 22 | 13 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2 | 7 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Axilla pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 9 | 2 | 4
Clavicular pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 2 | 0
Head soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Hip pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Jaw pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Knee pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 1 | 0
Muscle weakness left sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 9 | 6 | 3
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteonecrosis of lunate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 6 | 8 | 4
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 8 | 7 | 3
Abdominal numbness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 6 | 9 | 3
Dysarthria (Nervous system disorders) | 1 | 0 | 9 | 7 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 3 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Facial drooping (Nervous system disorders) | 0 | 0 | 0 | 3 | 0
Facial palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 9 | 6 | 3
Hypersomnia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Movements involuntary (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3 | 7 | 5 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 3 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 3 | 2
Confusion (Psychiatric disorders) | 0 | 0 | 7 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 3 | 4 | 1
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0 | 9 | 4 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 7 | 2 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 1
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 10 | 11 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 19 | 10 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 5 | 3
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 7 | 4 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Left vocal cord paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 6 | 3 | 3
Nasal regurgitation of liquids (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Oromaxillary fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 3 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 13 | 6 | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 7 | 3 | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 8 | 5 | 2
Bed sores (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Blisters on palms and toe (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermal neck nodules (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 18 | 11 | 10
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 7 | 3 | 0
Increased mucous secretions (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Lesion (unknown/furuncle) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 5 | 21 | 15 | 20
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 3 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 10 | 6 | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hematoma (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 2 | 4 | 25 | 13 | 12
Hypotension (Vascular disorders) | 0 | 0 | 7 | 5 | 2
Lymphedema (Vascular disorders) | 0 | 0 | 4 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT02101034/Prot_SAP_000.pdf